CLINICAL TRIAL: NCT01315444
Title: Gradual Cessation of Proton Pump Inhibitor (PPI) Treatment May Prevent Rebound Acid Secretion in Dyspeptic and Reflux Patients, Measured by the Alkaline Tide Method.
Brief Title: Gastric Acid Rebound Secretion Measured by Alkaline Tide
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Yaron Niv, Director, Department of Gastroenterology, Tel Aviv University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AT 101; RMC 101 (Other: RMC 101)
Record Dates: First submitted 2011-03-13; First posted 2011-03-15 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Condition Measuring Alkaline Tide and Filling Symptoms' Questionnaire After Abrupt or Gradual Step Down Cessation of PPI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPI abrupt cessation (Active Comparator): Abrupt cessation
  Interventions: Drug: Stop PPI gradually
- PPI gradual step down cessation (Active Comparator): Gradual cessation
  Interventions: Drug: Stop PPI gradually

INTERVENTIONS:
Drug: Stop PPI gradually
  Arms: PPI abrupt cessation
Drug: Stop PPI gradually
  Arms: PPI gradual step down cessation

SUMMARY:
Gastro esophageal reflux disease and ulcer related or non-ulcer dyspepsia, attacks 20% of the Western population. These millions of patients are treated continuously with PPI for different periods, many for many years. Recently, rebound acid hypersecretion was recognized as a major clinical event after cessation of PPI therapy. Sustained hypergastrinemia due to daily PPI therapy causes increased acid-secretory capacity that appears when the drug is stopped. The transient increase in blood and urinary pH following gastric secretion has been termed the alkaline tide phenomenon. Carbonic acid, formed in the presence of the enzyme carbonic anhydrase, neutralizes intracellular hydroxyl ions produced as a result of luminal acid secretion. The bicarbonate generated is removed from the cell via the baso-lateral chloride bicarbonate exchanger. The investigators have shown in several studies that this phenomenon parallels acid secretion. Thus, stimulation of acid secretion with test meal increased base excess maximally after 45 minutes and these changes parallel peak acid output measured in gastric aspirate. The investigators hypothesize that gradual step down cessation of PPI will prevent this clinical relevant event. By measuring alkaline tide after PPI cessation the investigators may prove this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Dyspepsia and reflux patients older than 18

Exclusion Criteria:

* patients on PPI, patients with severe diseases, younger than 18 y, older than 80 y, un-cooperative, COPD, uncompensated IHD, CRF

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
prevention of acid rebound phenomenon after stoping PPI | 30 days
  Comparing gradual and abrupt PPI cesation